CLINICAL TRIAL: NCT02895243
Title: Prehabilitation for Adults With End Stage Renal Disease on the Kidney Transplant Waitlist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00006786
Record Dates: First submitted 2016-09-06; First posted 2016-09-09 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Preoperative Exercise; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prehabilitation (Experimental)
  Interventions: Other: Prehabilitation

INTERVENTIONS:
Other: Prehabilitation — The study will use a generic prehabilitation program which will include the following components: Warm-up, cardiovascular training, strength training, flexibility training, and cool down. Prehabilitation will occur once per week and approximately 1 hour in duration. Participants will take part in prehabilitation until they receive a kidney transplant which by study design is approximately for 3-6 months.
  Other Names: exercise training

SUMMARY:
This pilot study will be a clinical trial to test the feasibility and effectiveness of a kidney transplant (KT) prehabilitation intervention in adults with end stage renal disease (ESRD) who are within 3-6 months of transplantation.

DETAILED DESCRIPTION:
Prehabilitation is the enhancement of functional capacity of a patient to improve their ability to withstand a future stressor. The investigators primary objective is to demonstrate feasibility for prehabilitation in Aim 1 and test whether the number of prehabilitation sessions is associated with increased physical activity. The investigators will formally test whether prehabilitation is associated with a reduction in short term and long term KT outcomes as part of Aim 2. The investigators will test whether there is an effect of prehabilitation on short-term (KT length of stay> 2 weeks, early hospital readmission and delayed graft function) and long-term (acute rejection (within the first year), 1 year patient and graft survival) outcomes compared to standard of care controls. Participants will be followed for 3-6 months or until they receive a kidney transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with end stage renal disease who are within 3-6 months of kidney transplantation and are on the kidney transplant waitlist at Johns Hopkins
2. Must be at least 18 years or older at enrollment
3. Must be English speaking
4. Must be enrolled in an ongoing cohort study of adults with ESRD who are being evaluated for kidney transplantation
5. Must be willing to participate in a prehabilitation program and able to give informed consent

Exclusion Criteria:

1. Patients who have any of the following medical conditions will be excluded from the study:

   * Active Angina pectoris
   * Chronic lung disease and daily use of oxygen
   * Cerebral vascular disease
   * Musculoskeletal conditions that would limit participation in prehabilitation
   * Lower- or upper-extremity amputation
   * Orthopedic disorders exacerbated by physical activity
   * Decreased mental capacity
2. Patients who live outside of Maryland will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Post kidney transplant mortality | 1 year
  1 year patient survival

CONTACTS AND LOCATIONS:
Overall Officials: Mara McAdams DeMarco, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Physical Medicine and Rehabilitation, Lutherville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No